CLINICAL TRIAL: NCT04807088
Title: Effect of Tactile-Kinesthetic Stimulation on Growth, Neurobehavior and Development Among Preterm Neonates
Brief Title: Effect of Tactile-Kinesthetic Stimulation on Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Prof. Hartono Gunardi, MD, PhD, Consultant Pediatrician, Head of Growth and Development-Social Pediatrics Division, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 681/UN2.F1/ETIK/2015
Record Dates: First submitted 2021-03-12; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Infant, Premature, Diseases
Keywords: preterm; growth; development; premature birth; infant; massage; weight gain
MeSH Terms: conditions — Infant, Premature, Diseases; Premature Birth; Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Tactile-kinesthetic stimulation (TKS) was performed with a specific baby oil provided by the investigator. Tactile stimulation was performed while the neonate was in prone position. Light massage was applied in the head, shoulder, back, legs and arms of the infants. Every massage was performed for 2 × 5 seconds, with a total duration of 5 minutes. Kinesthetic stimulation, including elbow flexion-extension movement, palm massages, flexion-extension of the knees and legs and plantar massages, was applied while the neonate was in supine position. Each kinesthetic stimulation was performed for 2 × 5 seconds. Each movement was repeated six times, with a total duration of 5 minutes. Tactile stimulation was repeated once after kinesthetic stimulation. The total duration of TKS was 15 minutes which was performed three times daily preferably between breastfeeding or bottle feeding for 10 consecutive days.
  Interventions: Procedure: Tactile-kinesthetic Stimulation
- Control Group (Placebo Comparator): Control group was not given TKS.
  Interventions: Other: Placebo

INTERVENTIONS:
Procedure: Tactile-kinesthetic Stimulation
  Arms: Intervention Group
Other: Placebo
  Arms: Control Group

SUMMARY:
An interventional study to evaluate the effect of tactile-kinesthetic stimulation (TKS) on growth, neurobehavior and development among preterm neonates in the neonatal unit of Dr. Cipto Mangunkusumo Hospital.

DETAILED DESCRIPTION:
Preterm neonates were recruited via random sampling and divided into two groups (intervention group and control group). A written informed consent was obtained from the parents or guardians.

Before the intervention, physical examination was performed to ensure the neonates had normal vital signs, were healthy and did not present with congenital abnormalities.

In the intervention group, TKS was performed with specific baby oil for 15 minutes, three times a day, for 10 days. After 10 days, TKS was applied once daily by the mother or caregiver. TKS implementation at home was supervised by the investigator or nurse through phone call. The TKS were documented by the mother or caregiver in the diary card, which should be brought during the next visit when the neonate was 11-14 days old. In addition to TKS, history of illness and nutrition which was confirmed through history taking during hospital or home visit, was also recorded. The participants who did not go the hospital were home visited by the investigator or nurse.

Anthropometric measurement by investigator and trained nurses and Dubowitz examination was performed by investigator in a warm and quiet place in the neonatal unit, mother-baby unit, outpatient clinic or participants' home while the neonate was fully alert.

At 3 months of age, infant development was assessed by the investigator using the Capute scales (Developmental Quotient of Clinical Adaptive Test [DQ CAT], Clinical Linguistic Adaptive Milestone Scale [DQ CLAMS]) and the Full Scale Developmental Quotient (FS DQ) score. The Clinical Linguistic Adaptive Milestone Scale (CLAMS) score was based on the parent's report of language skill attainment. The Clinical Adaptive Test (CAT) score was based on the child's performance according to the listed items.

ELIGIBILITY:
Inclusion Criteria:

* 6-24-hour-old preterm infants with 32-<37 gestational weeks
* birth weight ranging from 1,500 to <2,500 g
* appropriate for gestational age
* a minimum Apgar score of seven at the fifth minute
* no history of neonatal resuscitation
* stable vital condition
* no invasive therapy during hospitalisation

Exclusion Criteria:

* intrauterine growth retardation
* untreated clinical sepsis
* congenital abnormalities such as congenital heart disease
* history of hyperbilirubinemia

Ages: 6 Hours to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Change from Birth Body Weight at 11 Days Old | On the first day and 11 days old.
  Scale in grams. Using calibrated baby scale with accuracy of 10g, plotted in 2013 Fenton growth chart. The measurement was obtained twice if the same result was obtained and three times if the results differed. The mean was calculated.
Change from Birth Body Weight at 40 Weeks of Postmenstrual Age | On the first day and 40 weeks of postmenstrual age.
  Scale in grams. Using calibrated baby scale with accuracy of 10g, plotted in 2013 Fenton growth chart. The measurement was obtained twice if the same result was obtained and three times if the results differed. The mean was calculated.
Change from Birth Body Weight at 3 Months Old | On the first day and 3 months old.
  Scale in grams. Using calibrated baby scale with accuracy of 10g, plotted in 2013 Fenton growth chart. The measurement was obtained twice if the same result was obtained and three times if the results differed. The mean was calculated.
Change from Birth Body Length at 11 Days Old | On the first day and 11 days old.
  Scale in centimeters. Using a length board, plotted in 2013 Fenton growth chart.
Change from Birth Body Length at 40 Weeks of Postmenstrual Age | On the first day and 40 weeks of postmenstrual age.
  Scale in centimeters. Using a length board, plotted in 2013 Fenton growth chart.
Change from Birth Body Length at 3 Months Old | On the first day and 3 months old.
  Scale in centimeters. Using a length board, plotted in 2013 Fenton growth chart.
Change from Birth Head Circumference at 11 Days Old | On the first day and 11 days old.
  Scale in centimeters. Using a non-elastic tape, plotted in 2013 Fenton growth chart. Head circumference was measured three times from the glabella to the posterior occiput, and the largest measurement was recorded.
Change from Birth Head Circumference at 40 Weeks of Postmenstrual Age | On the first day and 40 weeks of postmenstrual age.
  Scale in centimeters. Using a non-elastic tape, plotted in 2013 Fenton growth chart. Head circumference was measured three times from the glabella to the posterior occiput, and the largest measurement was recorded.
Change from Birth Head Circumference at 3 Months Old | On the first day and 3 months old.
  Scale in centimeters. Using a non-elastic tape, plotted in 2013 Fenton growth chart. Head circumference was measured three times from the glabella to the posterior occiput, and the largest measurement was recorded.
Change from 6-24 hours of Age Neurobehavior at 11-14 Days of Age | 6-24 hours of age and 11-14 days of age.
  Using Dubowitz examination. The minimum Dubowitz score is 0 and the maximum is 72.
Change from 6-24 hours of age Neurobehavior at Term or 40 Weeks of Postmenstrual Age | 6-24 hours of age and term or 40 weeks of postmenstrual age.
  Using Dubowitz examination. The minimum Dubowitz score is 0 and the maximum is 72.
Change from 6-24 hours of age Neurobehavior at 3 Months Old | 6-24 hours of age and 3 Months Old.
  Using Dubowitz examination. The minimum Dubowitz score is 0 and the maximum is 72.
Infant Development | 3 months of age.
  Using Capute scales.

CONTACTS AND LOCATIONS:
Overall Officials: Hartono Gunardi, MD, PhD, Principal Investigator — Pediatric Consultant, Head of Growth and Development-Social Pediatrics Division
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aliabadi F, Askary RK. Effects of tactile-kinesthetic stimulation on low birth weight neonates. Iran J Pediatr. 2013 Jun;23(3):289-94. PMID 23795251
- [Background] Alvarez MJ, Fernandez D, Gomez-Salgado J, Rodriguez-Gonzalez D, Roson M, Lapena S. The effects of massage therapy in hospitalized preterm neonates: A systematic review. Int J Nurs Stud. 2017 Apr;69:119-136. doi: 10.1016/j.ijnurstu.2017.02.009. Epub 2017 Feb 14. PMID 28235686
- [Background] Blencowe H, Cousens S, Chou D, Oestergaard M, Say L, Moller AB, Kinney M, Lawn J; Born Too Soon Preterm Birth Action Group. Born too soon: the global epidemiology of 15 million preterm births. Reprod Health. 2013;10 Suppl 1(Suppl 1):S2. doi: 10.1186/1742-4755-10-S1-S2. Epub 2013 Nov 15. PMID 24625129
- [Background] Diego MA, Field T, Hernandez-Reif M. Preterm infant weight gain is increased by massage therapy and exercise via different underlying mechanisms. Early Hum Dev. 2014 Mar;90(3):137-40. doi: 10.1016/j.earlhumdev.2014.01.009. Epub 2014 Jan 27. PMID 24480603
- [Background] Dosman CF, Andrews D, Goulden KJ. Evidence-based milestone ages as a framework for developmental surveillance. Paediatr Child Health. 2012 Dec;17(10):561-8. doi: 10.1093/pch/17.10.561. PMID 24294064
- [Background] Dubowitz L, Ricciw D, Mercuri E. The Dubowitz neurological examination of the full-term newborn. Ment Retard Dev Disabil Res Rev. 2005;11(1):52-60. doi: 10.1002/mrdd.20048. PMID 15856443
- [Background] Elmoneim MA, Mohamed HA, Awad A, El-Hawary A, Salem N, El Helaly R, Nasef N, Abdel-Hady H. Effect of tactile/kinesthetic massage therapy on growth and body composition of preterm infants. Eur J Pediatr. 2021 Jan;180(1):207-215. doi: 10.1007/s00431-020-03738-w. Epub 2020 Jul 14. PMID 32666281
- [Background] Akhavan Karbasi S, Golestan M, Fallah R, Golshan M, Dehghan Z. Effect of body massage on increase of low birth weight neonates growth parameters: A randomized clinical trial. Iran J Reprod Med. 2013 Jul;11(7):583-8. PMID 24639794
- [Background] Kulkarni A, Kaushik JS, Gupta P, Sharma H, Agrawal RK. Massage and touch therapy in neonates: the current evidence. Indian Pediatr. 2010 Sep;47(9):771-6. PMID 21048258
- [Background] Mathai S, Fernandez A, Mondkar J, Kanbur W. Effects of tactile-kinesthetic stimulation in preterms: a controlled trial. Indian Pediatr. 2001 Oct;38(10):1091-8. PMID 11677298
- [Background] Moddemann D, Shea S. The developmental paediatrician and neonatal follow-up. Paediatr Child Health. 2006 May;11(5):295. PMID 19030294
- [Background] Orton J, Spittle A, Doyle L, Anderson P, Boyd R. Do early intervention programmes improve cognitive and motor outcomes for preterm infants after discharge? A systematic review. Dev Med Child Neurol. 2009 Nov;51(11):851-9. doi: 10.1111/j.1469-8749.2009.03414.x. Epub 2009 Sep 1. PMID 19732117
- [Background] Sankaranarayanan K, Mondkar JA, Chauhan MM, Mascarenhas BM, Mainkar AR, Salvi RY. Oil massage in neonates: an open randomized controlled study of coconut versus mineral oil. Indian Pediatr. 2005 Sep;42(9):877-84. PMID 16208048
- [Background] Santos IS, Matijasevich A, Domingues MR, Barros AJ, Victora CG, Barros FC. Late preterm birth is a risk factor for growth faltering in early childhood: a cohort study. BMC Pediatr. 2009 Nov 16;9:71. doi: 10.1186/1471-2431-9-71. PMID 19917121
- [Background] Soriano CR, Martinez FE, Jorge SM. Cutaneous application of vegetable oil as a coadjutant in the nutritional management of preterm infants. J Pediatr Gastroenterol Nutr. 2000 Oct;31(4):387-90. doi: 10.1097/00005176-200010000-00011. PMID 11045835
- [Background] Vickers A, Ohlsson A, Lacy JB, Horsley A. Massage for promoting growth and development of preterm and/or low birth-weight infants. Cochrane Database Syst Rev. 2004;2004(2):CD000390. doi: 10.1002/14651858.CD000390.pub2. PMID 15106151
- [Background] Woythaler MA, McCormick MC, Smith VC. Late preterm infants have worse 24-month neurodevelopmental outcomes than term infants. Pediatrics. 2011 Mar;127(3):e622-9. doi: 10.1542/peds.2009-3598. Epub 2011 Feb 14. PMID 21321024